CLINICAL TRIAL: NCT05216250
Title: A Phase 2 Multicenter, Randomized, Double-blind, Placebo-controlled Study of BOTOX® (Botulinum Toxin Type A) Purified Neurotoxin Complex for the Treatment of Upper Limb Essential Tremor
Brief Title: Study of BOTOX Injections to Assess Change in Disease Symptoms in Adult Participants With Upper Limb Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: M21-471; 2021-002191-39 (EudraCT Number)
Record Dates: First submitted 2021-10-01; First posted 2022-01-31 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Upper Limb Essential Tremor (UL ET)
Keywords: Upper Limb Essential Tremor; UL ET; BOTOX; Botulinum Toxin Type A
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- BOTOX/BOTOX Unilateral (Experimental): Participants will receive BOTOX in Cycle 1 and Cycle 2 and unilateral BOTOX in Cycle 3
  Interventions: Biological: BOTOX
- BOTOX/BOTOX Bilateral (Experimental): Participants will receive BOTOX in Cycle 1 and Cycle 2 and bilateral BOTOX in Cycle 3
  Interventions: Biological: BOTOX
- Placebo/BOTOX Unilateral (Experimental): Participants will receive placebo in Cycle 1 and Cycle 2 followed by unilateral BOTOX in Cycle 3.
  Interventions: Biological: BOTOX; Drug: Placebo for BOTOX
- Placebo/BOTOX Bilateral (Experimental): Participants will receive placebo in Cycle 1 and Cycle 2 followed by bilateral BOTOX in Cycle 3.
  Interventions: Biological: BOTOX; Drug: Placebo for BOTOX

INTERVENTIONS:
Biological: BOTOX — Intramuscular injection
  Other Names: Botulinum Toxin Type A
Drug: Placebo for BOTOX — Intramuscular injection
  Arms: Placebo/BOTOX Bilateral; Placebo/BOTOX Unilateral

SUMMARY:
Upper limb essential tremor (UL ET) is a movement disorder characterized by postural and/or kinetic tremor. It can cause difficulty with everyday tasks such as writing, pouring, and eating, and patients also experience associated social embarrassment. This study will assess how safe and effective BOTOX is in treating UL ET. Adverse events and change in disease activity will be evaluated.

BOTOX is an investigational drug being developed for the treatment of UL ET. Participants are randomly assigned to 1 of the 4 groups, called treatment arms. Each group receives different treatment. There is 1 in 2 chance that participants will be assigned to placebo. Around 174 participants, aged 18 to 80 years with UL ET will be enrolled in approximately 40 sites in North America.

Participants will receive BOTOX or placebo injections in Cycle 1 and Cycle 2. In Cycle 3, participants will receive unilateral or bilateral BOTOX injections. Each cycle is 12 weeks.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of essential tremor in accordance with modified Tremor Investigation Group (TRIG) criteria as described in the protocol.
* TREDS-Revised Scale (1-4 scale, whole numbers) unilateral score of >= 3 for the Tremor Disability Scale (TREDS) on any of the 7 unilateral items; no more than a single item score of 1 among the 7 unilateral items in the dominant limb.
* TETRAS activities of daily living (ADL) (recorded on a 0-4 scale, whole numbers) minimum score of >= 3 on any of the 5 unilateral items; no more than a single item score of <=1 among the 5 unilateral items in the dominant limb.
* At least one of the following criteria must also be met:

  * TETRAS UL score (0-4 scale, with 0.5 increments) of > 2 in the dominant limb on at least one of the 3 maneuvers OR
  * TETRAS Archimedes spiral task score (0-4 scale, with 0.5 increments) of > 2 in the dominant limb

Exclusion Criteria:

* Any uncontrolled clinically significant medical condition other than the one under study.
* Any medical condition that may put the participant at increased risk with exposure to BOTOX Purified Neurotoxin Complex.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2022-04-12 (Actual); Primary Completion 2025-02-03 (Actual); Study Completion 2025-02-03 (Actual)

PRIMARY OUTCOMES:
Change From Baseline in Tremor Disability Scale-Revised (TREDS-R) Total Score Across 7 Unilateral Items | Week 24
  Tremor Disability Scale-Revised (TREDS-R) is a scale to assess activities of daily living (ADL) through a self-questionnaire asking participants to rate how easy or difficult it is to perform a particular activity. The scale consists of 20 items with each item rated on a scale of 1 (able to do the activity without difficulty) to 4 (cannot do the activity by yourself). 7 items included in this subset will be: use a spoon to drink soup, hold a cup of tea, pour milk from a bottle or carton, dial a telephone, pick up your change in a shop, insert an electric plug into a socket, unlock your front door with a key.
Number of Participants with Treatment Emergent Adverse Events (AEs) | Up to approximately 36 weeks
  An AE is defined as any untoward medical occurrence in a patient or clinical investigation in which a participant is administered a pharmaceutical product which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Change From Baseline in TETRAS Activity of Daily Living (TETRAS ADL) Total Score Across 5 Unilateral Items | Week 24
  TETRAS Activity of Daily Living (TETRAS ADL) is a clinical rating scale using the total score across 5 unilateral items of the analyzed 10-item TETRAS ADL, with each item's recorded scores of 0 and 1 (0-4 scale) combined into one category with a score of 1 for analysis on a 1-4 scale.
  The 5 tasks included in this subset will be feeding with a spoon, drinking from a glass, pouring, using keys, and writing.
Change From Baseline in TETRAS Archimedes Spiral Score | Week 24
  Tremor Research Group Essential Tremor Rating Assessment Scale (TETRAS) Archimedes Spiral is an item of the TETRAS performance subscale that is designed to assess tremor severity. During this test, participants are instructed to draw an unbroken spiral which is then scored from 0 to 4, with 1 being tremor is "barely visible" and 4 being "figure not recognizable."
Change From Baseline in TETRAS Handwriting Score | Week 24
  TETRAS Handwriting is an item of the TETRAS performance subscale that is designed to assess tremor severity. During this test, participants are instructed to write the standard sentence "This is a sample of my best handwriting" using the dominant hand only, which is then scored from 0 to 4 with 1 being tremor is "slight: untidy due to tremor that is barely visible" and 4 being "severe: completely illegible."
Change From Baseline in Clinical Global Impression of Severity (CGI-S) | Week 24
  CGI-S is a single item used to measure the clinician's impression of the current severity of the patient's essential tremor. The measure uses a 5-point rating scale where "0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe."
Change From Baseline in Patient Global Impression of Severity (PGI-S) | Week 24
  PGI-S is a single item used to measure the participant's impression of severity of their essential tremor symptoms. The measure uses a 5-point rating scale where 0 = none, 1 = mild, 2 = moderate, 3 = severe, and 4 = very severe.
Change From Baseline in Essential Tremor Rating Assessment (TETRAS UL) Score | Week 24
  TETRAS Upper Limb (UL) Scale is an item of the TETRAS performance subscale that is designed to assess upper limb tremor during three maneuvers: forward horizontal reach posture, lateral "wing beating" posture, and finger-nose-finger testing. Each maneuver is scored from 0 to 4, with 1 indicating a tremor amplitude that is "barely visible" and 4 indicating a tremor amplitude that is >= 20 cm.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (40):
- United States (36):
  - Accel Research Sites - Neurology and Neurodiagnostics of Alabama, LLC /ID# 240472, Hoover, Alabama
  - Barrow Neurological Institute - Dignity Health St. Joseph's Hosp and Medical Ctr /ID# 231731, Phoenix, Arizona
  - University of Arizona /ID# 239781, Tucson, Arizona
  - Loma Linda University /ID# 230905, Loma Linda, California
  - University of Colorado - Anschutz Medical Campus /ID# 239869, Aurora, Colorado
  - New England Institute for Clinical Research /ID# 238404, Stamford, Connecticut
  - Parkinson's Disease and Movement Disorders Center of Boca Raton /ID# 231677, Boca Raton, Florida
  - Coastal Clinical Research Specialists /ID# 240897, Fernandina Beach, Florida
  - Coastal Clinical Research Specialists /ID# 240471, Jacksonville, Florida
  - Charter Research - Winter Park /ID# 241568, Orlando, Florida
  - CDC Research Institute LLC /ID# 242744, Port Saint Lucie, Florida
  - Emory University / Emory Brain Health Center /ID# 231911, Atlanta, Georgia
  - Accel Research Site-NeuroStudies /ID# 239881, Decatur, Georgia
  - Univ Kansas Med Ctr /ID# 231166, Kansas City, Kansas
  - Kansas Institute of Research /ID# 231623, Overland Park, Kansas
  - Tufts Medical Center /ID# 239929, Boston, Massachusetts
  - Lahey Hospital & Medical Center /ID# 233232, Burlington, Massachusetts
  - Henry Ford Health Medical Center - Jackson /ID# 231400, Jackson, Michigan
  - Dent Neurologic Institute - Amherst /ID# 255665, Amherst, New York
  - UNC Hospitals Neurology Clinic - Chapel Hill /ID# 238857, Chapel Hill, North Carolina
  - Neurology - Triad /ID# 239806, Winston-Salem, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 233550, Winston-Salem, North Carolina
  - Dayton Center for Neurological Disorders /ID# 233737, Centerville, Ohio
  - The Orthopedic Foundation /ID# 232234, New Albany, Ohio
  - Oregon Health and Science University /ID# 231581, Portland, Oregon
  - Thomas Jefferson University Hospital /ID# 232614, Philadelphia, Pennsylvania
  - University of Pittsburgh MC /ID# 233735, Pittsburgh, Pennsylvania
  - Medical University of South Carolina /ID# 233538, Charleston, South Carolina
  - Texas Neurology /ID# 250428, Dallas, Texas
  - University of Texas Southwestern Medical Center /ID# 239770, Dallas, Texas
  - Texas Movement Disorder Specialists, PLLC /ID# 242524, Georgetown, Texas
  - Baylor College of Medicine /ID# 231624, Houston, Texas
  - Univ Texas HSC San Antonio /ID# 232615, San Antonio, Texas
  - Integrated Neurology Services - Falls Church /ID# 233545, Falls Church, Virginia
  - Gamma Therapeutic Center /ID# 232547, Greenfield, Wisconsin
  - Marshfield Clinic - Marshfield /ID# 233191, Marshfield, Wisconsin
- Canada (4):
  - Vancouver Coastal Health Authority - University of British Columbia /ID# 240356, Vancouver, British Columbia
  - Centricity Research /ID# 240587, Halifax, Nova Scotia
  - Toronto Western Hospital /ID# 231587, Toronto, Ontario
  - Genge Partners /ID# 251546, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing, please refer to the link below.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Use Agreement (DUA). For more information on the process, or to submit a request, visit the following link.
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M21-471